CLINICAL TRIAL: NCT03834467
Title: Testing a Shortened Version of the AlAn's Game, Which Can be Delivered Through REDCap, in a Sample of Emerging Adults
Brief Title: Testing a Shortened Version of the AlAn's Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-0182
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Psychopathic Personality Trait
Keywords: psychopathic traits; moral elevation; prosocial behavior
MeSH Terms: conditions — Altruism

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned to receive one of two possible orders of administration. All subjects will first complete the Levenson Psychopathy Scale. Then Arm 1 presents the Moral Elevation stimulus after playing the first AlAn's Short Game v.2 (session 1), while Arm 2 presents the control stimulus (nature video). Subjects in both arms will then play AlAn's game again. After playing the game for a second time, subjects in both arms will fill out an Adverse Childhood Experiences Questionnaire (ACES), Social Connectedness survey, and Demographics form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Elevation Stimulus Video (Experimental): All subjects complete the Levenson Psychopathy Scale first. Arm 1 then presents the Moral Elevation stimulus video after playing the first AlAn's Short Game v.2 (session 1). Participants will then play the AlAn's Short Game v.2 (session 2) for a second time and then fill out an Adverse Childhood Experiences Questionnaire (ACES), Social Connectedness survey, and Demographics form.
  Interventions: Other: Arm 1 - Elevation Stimulus Video
- Arm 2 - Control Stimulus Video (Sham Comparator): All subjects complete the Levenson Psychopathy Scale first. Arm 2 then presents the control stimulus (nature video) after playing the first AlAn's Short Game v.2 (session 1). Participants will then play the AlAn's Short Game v.2 (session 2) for a second time and then fill out an Adverse Childhood Experiences Questionnaire (ACES), Social Connectedness survey, and Demographics form.
  Interventions: Other: Arm 2 - Control Stimulus Video

INTERVENTIONS:
Other: Arm 1 - Elevation Stimulus Video — Subjects will watch a video that has been shown in previous studies to elicit an elevation response. This video shows a news story about a man saving the life of another man who falls onto the subway tracks.
  Arms: Arm 1 - Elevation Stimulus Video
Other: Arm 2 - Control Stimulus Video — Subjects will watch a nature video.
  Arms: Arm 2 - Control Stimulus Video

SUMMARY:
It has been demonstrated that behavior on the AlAn's (altruism-antisocial) game is related to Moral Elevation response. Moral Elevation is a positive response to another's act of generosity "of charity, gratitude, fidelity, generosity or any other strong display of virtue". The constellation of emotional, physical and psychological aspects of a Moral Elevation response have been well described. Moral Elevation can be elicited with stimulus stories or videos and measured with self-report questionnaires. The experience of Moral Elevation is associated with subsequent prosocial and affiliative behaviors. Additionally, the research has linked Moral Elevation response with behavior on the AlAn's game. This study will test whether behavior on the AlAn's Short Game v.2 is related to Moral Elevation response and extend prior work by testing whether viewing the Moral Elevation stimulus prior to playing the AlAn's Short Game v.2 is associated with differences in game behavior. The study will also test whether psychopathic traits will correlate with game behavior.

DETAILED DESCRIPTION:
Hypotheses and Specific Aims:

Aim 1: Examine the similarities and differences in behaviors on the AlAn's Short Game v.2 seen with the two Active Trial (AT) types (where Red Cross donation will be reduced and subject will gain money (AT1) vs. where the Red Cross donation will increase and study participants will lose money (AT2).

Hypothesis 1: Number of accepted trials of AT1 and AT2 from session 1 will significantly correlate.

Aim 2: Test the effects of Elevation vs. Nature video on change in AlAn's Short Game v.2 behavior between sessions 1 and 2.

Hypothesis 2: Subjects who view the Elevation stimulus video (study Arm 1) will show increases in prosocial behavior while those watching the Nature video will not.

Aim 3: Test the association between psychopathic traits and Costly Helping and determine whether the influence of Elevation on Costly Helping dissipates with increasing levels of psychopathic traits.

Hypothesis 3: Psychopathic traits, as measured by the Levenson Self Report Psychopathy Scale, will significantly and negatively correlate with the amount of prosocial behavior in session 1.

Hypothesis 4: Using subjects from study Arm 1, change in AlAn's Short game v.2 behavior (session 2 minus session 1) will be negatively correlated with psychopathic trait scores.

ELIGIBILITY:
Inclusion Criteria:

• age 18-25 years

Exclusion Criteria:

• refusal to provide informed consent

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 537 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2019-10-26 (Actual); Study Completion 2019-10-26 (Actual)

PRIMARY OUTCOMES:
Change in the Amount of Prosocial Behavior on the AlAn's Short Game v.2 | within 45 minutes, during one single study visit
  The primary outcome of interest is the change in the amount of prosocial behavior on the AlAn's Short game between sessions 1 and 2 (Costly Helping session 2 minus Costly Helping session 1).
  Our two main analyses of interest using this outcome measure are: (1) to test whether viewing the Moral Elevation stimulus video vs. the Control video experience a greater change in Costly Helping (e.g., that Moral Elevation response promotes prosocial behavior); and (2) to test whether psychopathic traits attenuate the relationship between Moral Elevation and prosocial behavior (i.e., among those viewing the Moral Elevation stimulus video, that our primary outcome - change in prosocial behavior - will be negatively related to level of psychopathic traits).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T Sakai, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data. We might print the results of this research study in relevant journals or share aggregate data on that does not identify subjects with qualified investigators or as a supplement as required by some journals. However, the names and any other identifying information of research subjects will always be kept confidential and will not be shared. The data that may be shared in this manner include gender, age, and race/ethnicity, as well as responses from the AlAn's Game v.2, Levenson Psychopathy Scale, adverse childhood experiences questionnaire and social connectedness survey.

REFERENCES:
- [Background] Algoe SB, Haidt J. Witnessing excellence in action: the 'other-praising' emotions of elevation, gratitude, and admiration. J Posit Psychol. 2009;4(2):105-127. doi: 10.1080/17439760802650519. PMID 19495425
- [Background] Haidt J. Elevation and the positive psychology of morality. In: Keyes C, Haidt, J., editor. Flourishing: Positive psychology and the life well-lived. Washington, DC: American Psychological Association 913-919, 2003.
- [Background] Sakai JT, Dalwani MS, Mikulich-Gilbertson SK, McWilliams SK, Raymond KM, Crowley TJ. A Behavioral Measure of Costly Helping: Replicating and Extending the Association with Callous Unemotional Traits in Male Adolescents. PLoS One. 2016 Mar 15;11(3):e0151678. doi: 10.1371/journal.pone.0151678. eCollection 2016. PMID 26977935
- [Background] Aquino K, McFerran B, Laven M. Moral identity and the experience of moral elevation in response to acts of uncommon goodness. J Pers Soc Psychol. 2011 Apr;100(4):703-18. doi: 10.1037/a0022540. PMID 21443375
- [Background] Freeman D, Aquino K, McFerran B. Overcoming beneficiary race as an impediment to charitable donations: social dominance orientation, the experience of moral elevation, and donation behavior. Pers Soc Psychol Bull. 2009 Jan;35(1):72-84. doi: 10.1177/0146167208325415. Epub 2008 Nov 18. PMID 19017786